CLINICAL TRIAL: NCT06243926
Title: Clinical Outcomes Following the Sperm Selection by Rheotaxis and Thermotaxis in In-Situ Hand-made Microfluidics of Fluidic Walls in the Same ICSI Plate: a Randomized Controlled Trial
Brief Title: Sperm Selection by Rheotaxis and Thermotaxis in In-Situ Handmade Microfluidics of Fluidic Walls in the Same ICSI Plate
Acronym: IS-MFluidics
Status: Recruiting | Type: Observational
Sponsor: CREA Medicina de la Reproducción SL (Other)
Responsible Party: Sponsor
Other Study IDs: e.23.I
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Intracytoplasmic Sperm Injection; Sperm; Microfluidics
Keywords: ICSI; Sperm Selection; Microfluidics; Assisted Reproduction Techniques
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic; Sperm Capacitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Density gradient centrifugation (DGC): DGC is a protocol to select sperm based on their density and isopycnic points. It is a conventional protocol commonly used in IVF laboratories.
  Interventions: Other: Sperm selection for ICSI
- In-Situ rheotaxis handmade microfluidics (isM): The isM is a novel protocol to select sperm for ICSI based on microfluidics and sperm guidance responses to rheotaxis and thermotaxis. The isM protocol proved its efficacy and effectivity for ICSI in previous proof of concept and non-inferiority studies, respectively.
  Interventions: Other: Sperm selection for ICSI

INTERVENTIONS:
Other: Sperm selection for ICSI — Sperm selection for ICSI is a critical step to ensure the use of viable and healthy sperm for fertilization in vitro. The goal is to choose a sperm that has the best chance of resulting in a successful pregnancy.
  Other Names: Sperm capacitation; Sperm sorting; Sperm separation; Sperm recovery

SUMMARY:
Microfluidics technologies are proving their capability to select suitable sperm for ICSI, especially those that take advantage of the rheotaxic properties of sperm migration. In contrast to other sperm preparation methods such as Wash-Swim-Up and Density- Gradients-Centrifugation (DGC), microfluidics disregards washing and centrifugation steps along the procedure. However, microfluidics devices are costly and likely to fail to select motile sperm in dispermic samples. The investigators have recently described a novel approach for sperm selection by In-Situ handmade rheotaxis microfluidics of fluidic walls in the same ICSI plate. This methodology integrates a swim-over based on horizontal migration with a positive rheotaxis zone. The present study aims to deliver an unbiased comparison between two sperm selection techniques: DGC and In-Situ handmade rheotaxis microfluidics of fluidic walls (isM).

DETAILED DESCRIPTION:
Microfluidics technologies stand as the latest sperm selection methodology for ICSI. Increasingly, publications show novel and ingenious microfluidics strategies to integrate sperm biomimicry during in vitro sperm selection while simplifying the IVF workflow. Microfluidics are time-efficient methods which reduce the risks associated with handling, gamete mix-up and ROS production. However, microfluidics devices are costly and likely to fail to select motile sperm in dispermic samples. Aiming to outline the application of microfluidics in ART, the investigators conceived a lab-on-a-chip approach for sperm selection by In-Situ rheotaxis handmade microfluidics of fluidic walls. This microfluidics system allows selecting sperm for ICSI in the same ICSI-dish. Thus, from a microvolume of the raw semen sample, only using microfluidics, disregarding centrifugation, washing, plasticware, other cells, products or materials, and using the same culture medium needed to prepare the rest of the ICSI plate.

A previous proof-of-concept study showed that this methodology efficiently selected suitable sperm for ICSI. The investigators also demonstrated that the microfluidic protocol effectively separates at least 20 progressive spermatozoa in less than 15 minutes in a clean microdroplet, free of any remaining seminal plasma. A subsequent non-inferiority study showed that the microfluidic method performs as well as density gradient centrifugation to achieve ICSI outcomes such as fertilization and day-5 blastocyst formation rate, proving that In-Situ handmade rheotaxis microfluidics of fluidic walls are also effective in supporting pre-implantation embryonic development in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ICSI
* Female age under 40 years old
* Number of mature oocytes (MII) upon oocyte retrieval ≥ 6
* Male age under 50 years old
* Total number of progressive sperm ≥ 1 million

Exclusion Criteria:

* Patients with surgically retrieved sperm for ICSI
* Cases using cryopreserved oocytes
* Cases using cryopreserved sperm

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female:
  Age from 18 to 39 years old Number of mature oocytes (MII) upon oocyte retrieval ≥ 6
  Male:
  Age from 18 to 49 years old Total number of progressive sperm ≥ 1 million
Study Population: Couples enrolled in our IVF program, who meet the inclusion/exclusion criteria described above
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Fertilization Rate (FR) | 16 to 20 hours post-ICSI (day 1)
  The proportion of two-pronuclei zygote divided by the total number of matured and microinjected oocytes (2pn/MII, %)
Day 5 usable blastocyst rate (D5UBR) | 108 to 113 hours post-ICSI (day 5)
  The proportion of embryos classified as blastocysts at day 5 of development, which has been transferred and/or cryopreserved.
Blastocyst quality grade | 108 to 113 hours post-ICSI (day 5)
  Blastocysts are categorized following the scale described by the Spanish Association of Reproduction Biology Studies (ASEBIR). The ASEBIR classification categorizes blastocysts based on their morphology into four groups: from A (highest, better outcome) to D (lowest, worse outcome).

SECONDARY OUTCOMES:
Morphokinetics profile (MK PNa) | from 16 to 20 hours post-ICSI (day 1)
  The proportion of embryos showing the appearance of pronuclei (PNa) out of the expected time frame.
Morphokinetics profile (MK PNf) | from 24 to 25 hours post-ICSI (day 1)
  The proportion of embryos showing the fading of pronuclei (PNf) out of the expected time frame.
Morphokinetics profile (MK t2) | from 24 to 28 hours post-ICSI (day 1)
  The proportion of embryos showing 2 cells (t2) out of the expected time frame.
Morphokinetics profile (MK t4) | from 37 to 41hours post-ICSI (day 2)
  The proportion of embryos showing 4 cells (t4) out of the expected time frame.
Morphokinetics profile (MK t8) | from 51 to 69 hours post-ICSI (day 3)
  The proportion of embryos showing 8 cells (t8) out of the expected time frame.
Morphokinetics profile (MK tM) | from 81 to 96 hours post-ICSI (day 4)
  The proportion of embryos with full cell compaction (morula; tM) out of the expected time frame.
Morphokinetics profile (MK tSB) | from 99 to 101 hours post-ICSI (day 5)
  The proportion of embryos starting to blastulate (tSB) out of the expected time frame.
Morphokinetics profile (MK tB) | from 108 to 113 hours post-ICSI (day 5)
  The proportion of embryos starting to blastulate (tB) out of the expected time frame.
Implantation Rate (IR) | 5 to 6 gestational weeks
  The proportion of embryos that were transferred that develop to a gestational sac
Ongoing clinical pregnancy Rate (OCP) | 6 to 8 gestational weeks
  The proportion of embryos that were transferred that develop at least to the stage of fetal heart activity

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ruiz-Jorro MD, MSc, PhD, Principal Investigator — CREA. Medicina de la Reproducción S.L.
Locations (1):
- CREA Medicina de la Reproducción, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No